CLINICAL TRIAL: NCT04653207
Title: The Dose Effects of Isomaltulose and Sucrose on Glycaemic and Insulinemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/00025
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes; Obesity; Pre Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Glucose Intolerance | interventions — Sucrose; isomaltulose

STUDY DESIGN:
Intervention Model Description: Randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control 1 (Other): Glucose 50g
  Interventions: Other: Glucose Solution 1
- Control 2 (Other): Glucose 50g
  Interventions: Other: Glucose Solution 2
- Control 3 (Other): Glucose 50g
  Interventions: Other: Glucose Solution 3
- Sucrose/Isomaltulose 100:0 (Experimental): A drink with 50g sucrose/isomaltulose 100:0
  Interventions: Other: Sucrose/Isomaltulose 100:0
- Sucrose/Isomaltulose 0:100 (Experimental): A drink with 50g sucrose/isomaltulose 0:100
  Interventions: Other: Sucrose/Isomaltulose 0:100
- Sucrose/Isomaltulose 50:50 (Experimental): A drink with 50g sucrose/isomaltulose 50:50
  Interventions: Other: Sucrose/Isomaltulose 50:50
- Sucrose/Isomaltulose 60:40 (Experimental): A drink with 50g sucrose/isomaltulose 60:40
  Interventions: Other: Sucrose/Isomaltulose 60:40
- Sucrose/Isomaltulose 70:30 (Experimental): A drink with 50g sucrose/isomaltulose 70:30
  Interventions: Other: Sucrose/Isomaltulose 70:30
- Sucrose/Isomaltulose 80:20 (Experimental): A drink with 50g sucrose/isomaltulose 80:20
  Interventions: Other: Sucrose/Isomaltulose 80:20

INTERVENTIONS:
Other: Glucose Solution 1 — 50g glucose dissolve in 300ml of water
  Arms: Control 1
Other: Glucose Solution 2 — 50g glucose dissolve in 300ml of water
  Arms: Control 2
Other: Glucose Solution 3 — 50g glucose dissolve in 300ml of water
  Arms: Control 3
Other: Sucrose/Isomaltulose 100:0 — 50g sucrose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 100:0
Other: Sucrose/Isomaltulose 0:100 — 50g isomaltulose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 0:100
Other: Sucrose/Isomaltulose 50:50 — 25g sucrose and 25g isomaltulose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 50:50
Other: Sucrose/Isomaltulose 60:40 — 30g sucrose and 20g isomaltulose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 60:40
Other: Sucrose/Isomaltulose 70:30 — 35g sucrose and 15g isomaltulose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 70:30
Other: Sucrose/Isomaltulose 80:20 — 40g sucrose and 10g isomaltulose dissolve in 300ml of water
  Arms: Sucrose/Isomaltulose 80:20

SUMMARY:
This study will determine the glycaemic and insulinaemic response and sensory profile of the drinks with various ratios sucrose:isomaltulose. The information will be useful for manufacturers of beverages to produce blood glucose friendlier drinks. The information will also be useful for dieticians and clinicians in recommending foods and drinks for people with diabetes. The information will also be useful to the public for making better food choices. The data will also provide insights on how the different ratios of sweeteners may affect glycaemic and insulinaemic indices (GI and II).

DETAILED DESCRIPTION:
The aim of the study is to determine the optimal mixture of sucrose with isomaltulose that will produce optimal reduction in glycaemia and an acceptable sensory profile. These will be assessed among three different ethnicities.The study will recruit a maximum of 60 healthy young (21-60 years old) males from three ethnicities (Malay, Indian, and Chinese). Each participant will take part in 9 separate test sessions on nonconsecutive days, and consume 3 reference control drinks and 6 different test drinks. On each of the test days, participants will consume either the reference drink (50g of anhydrous glucose dissolved in 300 ml of water) or one of the test drinks which consists of 50g of sucrose and/or isomaltulose dissolved in 300 ml of water in the following ratios: 0:100, 100:0, 50:50, 80:20, 70:30, 60:40 sucrose:isomaltulose. Study population: The study will recruit a maximum of 65 healthy young (21-60 years old) males. At least 10 participants will be selected from the three ethnicities (Malay, Indian, and Chinese). Males will be selected in order to avoid effects of the menstrual cycle. Participants will be recruited from the general public in Singapore and will be between 21 and 60 years, with a body mass index between 22 and 27 kg/m2.Design: The experimental protocol adopted is a pre-validated method used repeatedly for measuring the GI of foods. The testing follows a randomised, single-blinded, between-subjects, crossover design with participants returning on 9 non-consecutive days. Reference food testing (standard glucose solution) will precede test food testing. On each test day, participant will consume either the reference drink or one of the test drinks. The test sessions will be made up of 3 identical reference drinks and 6 test drinks. The number sessions each participant will complete will be determined by the researcher and communicated to the participant. For the 9 test sessions, participants arrive at the laboratory between 8:30-9 am following a 10 hour overnight fast. They are instructed not to partake in intense level sports and avoid alcohol consumption on the evening prior to a test session. Following a 10 minute rest two blood samples are obtained five minutes apart for determining baseline blood glucose levels. They are then given either the standard or test drink to consume. They are instructed to consume the food at a comfortable pace within 12 minutes. After consumption of the test drink, subjects will complete a liking questionnaire. Further blood samples are obtained at 15, 30, 45, 60, 90, 120, 150 and 180 minutes for blood glucose measurements and insulin (at every half hour intervals).Reference/Test foods: The reference drink will be anhydrous glucose (50 g) (standard) dissolved in 300 ml of water) and will be consumed on 3 occasions. The test drinks will consist of 50g of sucrose and/or isomaltulose dissolved in 300 ml of water in the following ratios: 0:100, 100:0, 50:50, 80:20, 70:30, 60:40 sucrose:isomaltulose. A total of 6 test drinks will be tested. The participant will be requested to finish both reference and test drink within 12min.Blood collection: Participants will be asked to attend the testing sessions after an overnight fast of ten to twelve hours. Two fasting blood samples will be collected by finger prick for glucose measurement and not more than 0.5ml finger prick blood sample will also be collected to measure baseline insulin. A drop of blood will be collected into a HemoCue® cuvette (Helsingborg, Sweden) for blood glucose analysis. In addition, not more than 0.5ml of finger prick blood will be collected for the analyses of plasma insulin concentrations. Participants will then consume the test meal within 12 minutes. Following this, approximately 5µl of blood samples will be collected at 15, 30, 45, 60, 90, 120, 150 and 180min for glucose measurements and not more than 0.5ml of blood samples will be collected at 30, 60, 90, 120, 150 and 180min for insulin measurements.'Liking' questionnaire: On the testing session days, participants will be asked to rate their 'liking' for the test meal. Participants will be rate their 'overall liking' for the test meal on a 100 mm Visual Analog Scale anchored with 'dislike extremely' (0 mm), 'neither like nor dislike' (50 mm) and 'like extremely' (100 mm) immediately after they consume the test meal.Screening: Potential participants will first attend a screening session for consenting and eligibility procedures. Participants will arrive in the morning following an overnight fast. During the screening, a questionnaire will have to be completed and anthropometry and blood pressure will be assessed. Screening questionnaire: The screening questionnaire will include contact information, demographic, general health details, and physical activity level. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes. Anthropometric measurements: Body weight and body composition will be measured using bioelectrical impedance analysis. Height will be measured using a stadiometer in order to calculate participants' BMI. Waist circumference will be measured at the minimum circumference between the iliac crest and the rib cage. Hip circumference will be measured at the maximum protuberance of the buttocks. Blood pressure will also be measured. Blood pressure: Blood pressure will be measured using an Omron blood pressure monitor (Model HEM-907) at baseline. Participants will be seated for five minutes before blood pressure is measured. Measurements will be taken in duplicate and the averaged results will be recorded.

ELIGIBILITY:
* Males
* Asian selected from the three ethnicities Malay, Indian and Chinese
* Age between 21-60 years
* Do not partake in sports at the competitive and/or endurance levels
* Body mass index between 22 to 27 kg/m2
* Normal blood pressure (<140/80 mmHg)
* Fasting blood glucose <6 mmol/L
* Do not have an ongoing infection or currently undergoing treatment at the time of screening
* Do not have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Do not have active Tuberculosis (TB) or currently receiving treatment for TB
* Not on any concurrent research study/trials
* Do not smoke
* Do not have any metabolic diseases (such as diabetes, hypertension etc)
* Do not have glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Not having medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Do not have intolerances or allergies to foods including the test foods and fructose
* Do not partake in sports at the competitive and/or endurance levels
* Do not intentionally restrict food intake
* Do not have an ongoing infection or currently undergoing treatment at the time of screening
* Do not have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Do not have active Tuberculosis (TB) or currently receiving treatment for TB
* Not on any concurrent research study/trials • Do not smoke• Do not have any metabolic diseases (such as diabetes, hypertension etc)
* Do not have glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Not having medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)• Do not have intolerances or allergies to foods including the test foods and fructose
* Do not partake in sports at the competitive and/or endurance levels
* Do not intentionally restrict food intake
* Not a team member of the study or is an immediate family member (Immediate family defined as a spouse, parent, child, or sibling, whether biological or legally adopted)

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All healthy male participants
Enrollment: 64 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose over 180 minutes period | 180 minutes
  Blood obtained through fingerprick, analysed using Hemocue analyser.

SECONDARY OUTCOMES:
Change in postprandial plasma insulin over 180 minutes period | 180 minutes
  Capillary plasma obtained through finger prick, analysed using Cobas analyser

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore